CLINICAL TRIAL: NCT04243564
Title: Comparison of the ProSeal Laryngeal Mask and I-gel as a Temporary Ventilatory Device Before Tracheal Intubation in Morbidly Obese Patients
Brief Title: Laryngeal Mask in Morbid Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Device (ProSeal Laryngeal Mask Airway) no longer available
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3793AO16
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2021-01

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Investigators hypothesize PLMA and I-gel are both effective as temporary ventilatory device in morbidly obese patients.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLMA (Active Comparator): The PLMA, a second generation gastric access SGD, is used as temporary ventilatory device before tracheal intubation. Performance is evaluated.
  Interventions: Device: Supraglottic device (SGD)
- I-gel (Active Comparator): The I-gel, a second generation gastric access SGD, is used as temporary ventilatory device before tracheal intubation. Performance is evaluated.
  Interventions: Device: Supraglottic device (SGD)

INTERVENTIONS:
Device: Supraglottic device (SGD) — Positioning of SGD as temporary ventilatory device before tracheal intubation

SUMMARY:
Investigators study the performance of both masks, Proseal Laryngeal Mask Airway (PLMA) and I-gel, as temporary ventilatory supraglottic airway devices (SGDs) before tracheal intubation in morbidly obese patients. Data are lacking in such population of patients

DETAILED DESCRIPTION:
The available data regarding SGDs in morbidly obese patients have focused mainly on PLMA. In general, SGDs have been successfully used as temporary ventilatory devices before laryngoscope-guided tracheal intubation, conduits for endotracheal tube insertion, and primary airway devices during surgery. Second-generation SGDs are preferred for both rescue airway and routine use, compared with first-generation, non-gastric access devices. Data on comparison PLMA vs. I-gel in morbidly obese patient are lacking.

The PLMA is a second generation gastric access SGD. PLMA is composed of an airway tube that connects to a mask which, after insertion through the patient's mouth and inflation of cuff, forms an airtight seal on top the glottis allowing a secure airway to be managed by a health care provider. PLMA can be autoclaved and reused many times. I-gel is a new type of single use, second generation, gastric access SGD and doesn't have an inflatable cuff. Because of its thermoplastic elastomer structure, it exactly adapts to the supraglottic tissue by binding with body temperature, thus minimising air leakage.

The aim of this study is to compare PLMA and I-gel regarding insertion success rate, the time of insertion, gastric access tube positioning, oropharyngeal leak pressure, assessment of position by fiberoptic, ventilatory parameters and hemodynamic, and complications for each device placed before tracheal intubation in morbidly obese patients.

This study is conducted at University Medical Hospital of Padova, with approval from Hospital research Ethical Committee and written informed consents from patients,. Patients are randomly allocated into 2 equal groups, according to the inclusion and exclusion criteria.

PLMA (n=35) in which PLMA is used for ventilation. I-gel (n=35) in which I-gel is used for ventilation.

I

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patients scheduled for elective bariatric surgery under general anesthesia

Exclusion Criteria:

* nonfasting; symptoms or endoscopic evidence of gastroesophageal reflux, of gastric ulcer, or oropharyngeal pathology; known or predicted difficult airway; allergy to anesthetic and nonsteroidal antiinflammatory drugs; or inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure (OLP) | Procedure (After correct placement of SGD)
  OLP is defined as the anesthesia circuit pressure at which a gas leak occurs around the SGD

SECONDARY OUTCOMES:
Time insertion | Procedure (Time from pick up to correct placement of SGD)
  Time for definitive placement of SGD
SGD placement | Procedure (From pick up to correct placement of SGD)
  Ease of insertion of the SGD
Gastric tube | Procedure (After correct placement of SGD)
  Ease of insertion of the gastric tube through the dedicated conduit
fiberoptic evaluation | Procedure (After correct placement of SGD and established ventilation)
  Fiberoptic evaluation of correct positioning through SGD
Leak fraction | Procedure (After correct placement of SGD and established ventilation)
  The leak fraction is defined as the leak volume divided by the inspired tidal volume.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Carron, MD, Principal Investigator — University of Padova
Locations (1):
- University Padiua Hospital, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gasteiger L, Brimacombe J, Perkhofer D, Kaufmann M, Keller C. Comparison of guided insertion of the LMA ProSeal vs the i-gel. Anaesthesia. 2010 Sep;65(9):913-6. doi: 10.1111/j.1365-2044.2010.06422.x. PMID 20645948
- [Result] Keller C, Brimacombe J, Kleinsasser A, Brimacombe L. The Laryngeal Mask Airway ProSeal(TM) as a temporary ventilatory device in grossly and morbidly obese patients before laryngoscope-guided tracheal intubation. Anesth Analg. 2002 Mar;94(3):737-40; table of contents. doi: 10.1097/00000539-200203000-00048. PMID 11867408
- [Result] Van Zundert TC, Brimacombe JR. Similar oropharyngeal leak pressures during anaesthesia with i-gel, LMA-ProSeal and LMA-Supreme Laryngeal Masks. Acta Anaesthesiol Belg. 2012;63(1):35-41. PMID 22783708
- [Result] Maitra S, Baidya DK, Arora MK, Bhattacharjee S, Khanna P. Laryngeal mask airway ProSeal provides higher oropharyngeal leak pressure than i-gel in adult patients under general anesthesia: a meta-analysis. J Clin Anesth. 2016 Sep;33:298-305. doi: 10.1016/j.jclinane.2016.04.020. Epub 2016 May 18. PMID 27555181